CLINICAL TRIAL: NCT02699450
Title: A Multiple-Center, Multiple-Dose, Randomized, Active Comparator-Controlled, Double-Masked, Parallel Group, 36-Week Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of RO6867461 Administered Intravitreally in Patients With Diabetic Macular Edema
Brief Title: A Study of Faricimab (RO6867461) in Participants With Center-Involving Diabetic Macular Edema
Acronym: BOULEVARD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP30099; RG7716 (Other: Roche theme number)
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — faricimab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: 0.3 mg Ranibizumab (Active Comparator): Participants will receive 0.3 milligrams (mg) ranibizumab every fourth week up to Week 20, for a total of 6 administrations, followed by an observational period up to Week 36. If a participant meets pre-specified criteria the participant will receive a single dose of 0.3 mg ranibizumab and exit the study.
  Interventions: Drug: Ranibizumab
- Arm B: 1.5 mg Faricimab (Experimental): Participants will receive 1.5 mg faricimab every fourth week up to Week 20, for a total of 6 administrations, followed by an observational period up to Week 36. If a participant meets pre-specified criteria the participant will receive a single dose of 0.3 mg ranibizumab and exit the study.
  Interventions: Drug: Faricimab
- Arm C: 6 mg Faricimab (Experimental): Participants will receive 6 mg faricimab every fourth week up to Week 20, for a total of 6 administrations, followed by an observational period up to Week 36. If a participant meets pre-specified criteria the participant will receive a single dose of 0.3 mg ranibizumab and exit the study.
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — Faricimab will be administered by IVT injection in the study eye.
  Other Names: RO6867461; RG7716
  Arms: Arm B: 1.5 mg Faricimab; Arm C: 6 mg Faricimab
Drug: Ranibizumab — Ranibizumab will be administered by IVT injection in the study eye.
  Other Names: Lucentis
  Arms: Arm A: 0.3 mg Ranibizumab

SUMMARY:
This is a multiple-center, multiple-dose, randomized, active comparator-controlled, double-masked, three parallel group, 36-week study in participants with center-involving diabetic macular edema (DME). Only one eye will be selected as the study eye. Where both eyes meet all eligibility criteria, the eye with the worse best corrected visual acuity (BCVA) will be defined as the study eye. The study will consist of a treatment period (20 weeks) and an observational period (up to 16 weeks). Treatment naive participants will be randomized in a 1:1:1 ratio to one of the Arms A, B and C, respectively. Participants previously treated with intravitreal (IVT) anti-vascular endothelial growth factor (VEGF) will be randomized in a 1:1 ratio to Arms A and C.

ELIGIBILITY:
Inclusion Criteria:

* Macular edema associated with diabetic retinopathy
* Decreased visual acuity attributable primarily to DME
* Diagnosis of diabetes mellitus

Exclusion Criteria:

* High risk proliferative diabetic retinopathy
* Cataract surgery within 3 months of Baseline, or any other previous intraocular surgery
* Uncontrolled glaucoma
* Current or history of ocular disease in the study eye other than DME
* Major illness or major surgical procedure within 1 month prior to Day 1
* Uncontrolled blood pressure
* Glycosylated hemoglobin (HbA1c) greater than (>) 12 percent (%) at screening
* Untreated diabetes mellitus or initiation of oral anti-diabetic medication or insulin within 4 months prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (60):
- United States (60):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - Retina Consultants of Orange County, Fullerton, California
  - United Med Res Inst, Inglewood, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Ophthalmic Clinical Trials San Diego, Oceanside, California
  - Southern CA Desert Retina Cons, Palm Desert, California
  - Retina Consultants, San Diego, Poway, California
  - Retinal Consultants Med Group, Sacramento, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Consultants of Southern, Colorado Springs, Colorado
  - Rand Eye, Deerfield Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Univ of Illinois at Chicago, Chicago, Illinois
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Illinois Retina Associates SC, Oak Park, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Wilmer Eye Institute, Baltimore, Maryland
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Vitreoretinal Surgery, Edina, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - Retina Center of New Jersey, Bloomfield, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - Capital Region Retina, Albany, New York
  - Opthalmic Consultants of LI, Lynbrook, New York
  - Retina Consultants of Western New York, Orchard Park, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Cleveland Clinic Foundation; Cole Eye Institute, Cleveland, Ohio
  - OSU Eye Physicians & Surgeons, Columbus, Ohio
  - Oregon Retina, LLP, Eugene, Oregon
  - Retina Northwest, Portland, Oregon
  - Palmetto Retina Center, Florence, South Carolina
  - Charleston Neuroscience Inst, Ladson, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC., Nashville, Tennessee
  - W Texas Retina Consultants PA, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Austin, Austin, Texas
  - Retina Specialists, DeSoto, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Med Center Ophthalmology Assoc, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Univ of Virginia Ophthalmology, Charlottesville, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
  - West Virginia University Eye Institute, Morgantown, West Virginia

REFERENCES:
- [Derived] Sahni J, Patel SS, Dugel PU, Khanani AM, Jhaveri CD, Wykoff CC, Hershberger VS, Pauly-Evers M, Sadikhov S, Szczesny P, Schwab D, Nogoceke E, Osborne A, Weikert R, Fauser S. Simultaneous Inhibition of Angiopoietin-2 and Vascular Endothelial Growth Factor-A with Faricimab in Diabetic Macular Edema: BOULEVARD Phase 2 Randomized Trial. Ophthalmology. 2019 Aug;126(8):1155-1170. doi: 10.1016/j.ophtha.2019.03.023. Epub 2019 Mar 21. PMID 30905643

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 229 patients were randomized, but two participants randomized to Arm C: 6 mg Faricimab were excluded from the analysis populations due to Good Clinical Practice (GCP) non-compliance at a single site.
Groups:
- Arm A: 0.3 mg Ranibizumab: Participants received 0.3 milligrams (mg) ranibizumab every fourth week up to Week 20, for a total of 6 administrations, followed by an observational period up to Week 36. If a participant met pre-specified criteria they received a single dose of 0.3 mg ranibizumab and exited the study.
- Arm B: 1.5 mg Faricimab: Participants received 1.5 mg faricimab every fourth week up to Week 20, for a total of 6 administrations, followed by an observational period up to Week 36. If a participant met pre-specified criteria they received a single dose of 0.3 mg ranibizumab and exited the study.
- Arm C: 6 mg Faricimab: Participants received 6 mg faricimab every fourth week up to Week 20, for a total of 6 administrations, followed by an observational period up to Week 36. If a participant met pre-specified criteria they received a single dose of 0.3 mg ranibizumab and exited the study.
Period: Overall Study
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Started (Intent-to-Treat (ITT) Population) | 90 | 55 | 82
Received at Least One Dose of Study Drug (Safety Population) | 89 | 55 | 80
Completed up to Week 24 | 81 | 53 | 73
Completed (Completed Study (per pre-specified criteria)) | 75 | 50 | 67
Not Completed | 15 | 5 | 15
Not completed — Death | 2 | 1 | 2
Not completed — Met Criteria for Study Exit | 0 | 0 | 1
Not completed — Protocol Violation | 4 | 3 | 5
Not completed — Lost to Follow-up | 3 | 0 | 5
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two participants randomized to Arm C: 6 mg Faricimab were excluded from the analysis populations due to Good Clinical Practice (GCP) non-compliance at a single site.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab | Total
Number analyzed (Participants) | 90 | 55 | 82 | 227
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Baseline characteristics were analyzed for all participants, treatment-naive participants, and previously treated participants.
  Years
    All Participants | 62.3 (9.2) | 61.5 (7.7) | 60.8 (9.2) | 61.6 (8.8)
    Treatment-Naive Participants: number analyzed (Participants) | 59 | 54 | 53 | 166
    Treatment-Naive Participants | 61.6 (9.5) | 61.4 (7.7) | 60.5 (9.1) | 61.2 (8.8)
    Previously Treated Participants: number analyzed (Participants) | 31 | 1 | 29 | 61
    Previously Treated Participants | 63.5 (8.7) | 63.0 (NA) — Standard deviation could not be calculated from data for a single participant. | 61.5 (9.5) | 62.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics were analyzed for all participants, treatment-naive participants, and previously treated participants.
  Participants
    All Participants: Female | 36 | 35 | 36 | 107
    All Participants: Male | 54 | 20 | 46 | 120
    Treatment-Naive Participants: number analyzed (Participants) | 59 | 54 | 53 | 166
    Treatment-Naive Participants: Female | 22 | 35 | 20 | 77
    Treatment-Naive Participants: Male | 37 | 19 | 33 | 89
    Previously Treated Participants: number analyzed (Participants) | 31 | 1 | 29 | 61
    Previously Treated Participants: Female | 14 | 0 | 16 | 30
    Previously Treated Participants: Male | 17 | 1 | 13 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics were analyzed for all participants, treatment-naive participants, and previously treated participants.
  Participants
    All Participants: Hispanic or Latino | 15 | 8 | 16 | 39
    All Participants: Not Hispanic or Latino | 74 | 47 | 66 | 187
    All Participants: Unknown or Not Reported | 1 | 0 | 0 | 1
    Treatment-Naive Participants: number analyzed (Participants) | 59 | 54 | 53 | 166
    Treatment-Naive Participants: Hispanic or Latino | 11 | 8 | 9 | 28
    Treatment-Naive Participants: Not Hispanic or Latino | 48 | 46 | 44 | 138
    Treatment-Naive Participants: Unknown or Not Reported | 0 | 0 | 0 | 0
    Previously Treated Participants: number analyzed (Participants) | 31 | 1 | 29 | 61
    Previously Treated Participants: Hispanic or Latino | 4 | 0 | 7 | 11
    Previously Treated Participants: Not Hispanic or Latino | 26 | 1 | 22 | 49
    Previously Treated Participants: Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics were analyzed for all participants, treatment-naive participants, and previously treated participants.
  Participants
    All Participants: American Indian or Alaska Native | 1 | 0 | 2 | 3
    All Participants: Asian | 0 | 0 | 1 | 1
    All Participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    All Participants: Black or African American | 17 | 11 | 14 | 42
    All Participants: White | 71 | 43 | 61 | 175
    All Participants: More than one race | 0 | 0 | 0 | 0
    All Participants: Unknown or Not Reported | 1 | 1 | 4 | 6
    Treatment-Naive Participants: number analyzed (Participants) | 59 | 54 | 53 | 166
    Treatment-Naive Participants: American Indian or Alaska Native | 0 | 0 | 2 | 2
    Treatment-Naive Participants: Asian | 0 | 0 | 1 | 1
    Treatment-Naive Participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Treatment-Naive Participants: Black or African American | 9 | 11 | 10 | 30
    Treatment-Naive Participants: White | 49 | 42 | 39 | 130
    Treatment-Naive Participants: More than one race | 0 | 0 | 0 | 0
    Treatment-Naive Participants: Unknown or Not Reported | 1 | 1 | 1 | 3
    Previously Treated Participants: number analyzed (Participants) | 31 | 1 | 29 | 61
    Previously Treated Participants: American Indian or Alaska Native | 1 | 0 | 0 | 1
    Previously Treated Participants: Asian | 0 | 0 | 0 | 0
    Previously Treated Participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Previously Treated Participants: Black or African American | 8 | 0 | 4 | 12
    Previously Treated Participants: White | 22 | 1 | 22 | 45
    Previously Treated Participants: More than one race | 0 | 0 | 0 | 0
    Previously Treated Participants: Unknown or Not Reported | 0 | 0 | 3 | 3
Anti-VEGF Treatment Experience Status (Treatment-Naive or Previously Treated) [Count of Participants; unit: Participants] — Approximately 210 participants were planned to be randomized to this study, including approximately 150 treatment-naive participants (1:1:1 to Arms A, B, and C) and approximately 60 participants (1:1 to Arms A and C) who had been previously treated with IVT anti-vascular endothelial growth factor (VEGF).
  Participants
    Treatment-Naive | 59 | 54 | 53 | 166
    Previously Treated | 31 | 1 | 29 | 61
Best Corrected Visual Acuity (BCVA) ETDRS Letter Score in the Study Eye at Baseline [Mean (Standard Deviation); unit: Score on a scale] — Population: Baseline characteristics were analyzed for all participants, treatment-naive participants, and previously treated participants. This analysis included participants who had received at least one dose of study drug and had non-missing assessments at baseline.
  Score on a scale
    All Participants: number analyzed (Participants) | 89 | 55 | 80 | 224
    All Participants | 61.51 (10.43) | 61.16 (11.12) | 59.48 (12.49) | 60.70 (11.36)
    Treatment-Naive Participants: number analyzed (Participants) | 58 | 54 | 51 | 163
    Treatment-Naive Participants | 61.24 (9.87) | 60.94 (11.11) | 60.00 (10.95) | 60.75 (10.58)
    Previously Treated Participants: number analyzed (Participants) | 31 | 1 | 29 | 61
    Previously Treated Participants | 62.00 (11.56) | 73.00 (NA) — Standard deviation could not be calculated from data for a single participant. | 58.55 (14.98) | 60.54 (13.31)
Previous Macular Laser Treatment Status [Count of Participants; unit: Participants] — Population: Baseline characteristics were analyzed for all participants, treatment-naive participants, and previously treated participants.
  Participants
    All Participants: Previous Macular Laser Treatment | 16 | 4 | 15 | 35
    All Participants: No Previous Macular Laser Treatment | 74 | 51 | 67 | 192
    Treatment-Naive Participants: number analyzed (Participants) | 59 | 54 | 53 | 166
    Treatment-Naive Participants: Previous Macular Laser Treatment | 6 | 4 | 3 | 13
    Treatment-Naive Participants: No Previous Macular Laser Treatment | 53 | 50 | 50 | 153
    Previously Treated Participants: number analyzed (Participants) | 31 | 1 | 29 | 61
    Previously Treated Participants: Previous Macular Laser Treatment | 10 | 0 | 12 | 22
    Previously Treated Participants: No Previous Macular Laser Treatment | 21 | 1 | 17 | 39
Mean Foveal Center Point Thickness at Baseline [Mean (Standard Deviation); unit: micrometers] — Foveal center point thickness (FCPT) is defined as the thickness from the inner limiting membrane to the retinal pigment epithelial at the horizontal slice closest to the center of the fovea. Foveal center point thickness was measured using spectral domain optical coherence tomography (SD-OCT). Population: Baseline characteristics were analyzed for all participants, treatment-naive participants, and previously treated participants. This analysis included participants who had received at least one dose of study drug and had non-missing assessments at baseline.
  micrometers
    All Participants: number analyzed (Participants) | 89 | 55 | 80 | 224
    All Participants | 459.88 (162.09) | 494.64 (200.51) | 440.50 (150.42) | 461.49 (168.97)
    Treatment-Naive Participants: number analyzed (Participants) | 58 | 54 | 51 | 163
    Treatment-Naive Participants | 464.19 (166.00) | 497.78 (201.02) | 456.70 (156.12) | 472.97 (175.37)
    Previously Treated Participants: number analyzed (Participants) | 31 | 1 | 29 | 61
    Previously Treated Participants | 451.82 (156.87) | 325.00 (NA) — Standard deviation could not be calculated from data for a single participant. | 412.02 (137.83) | 430.82 (147.49)
Mean Central Subfield Thickness at Baseline [Mean (Standard Deviation); unit: micrometers] — Central subfield thickness (CST) is defined as the mean thickness from the inner limiting membrane to the retinal pigment epithelial over the 1 millimetre (mm) central subfield. Central subfield thickness was measured using SD-OCT. Population: Baseline characteristics were analyzed for all participants, treatment-naive participants, and previously treated participants. This analysis included participants who had received at least one dose of study drug and had non-missing assessments at baseline.
  micrometers
    All Participants: number analyzed (Participants) | 89 | 55 | 80 | 224
    All Participants | 489.01 (136.74) | 532.89 (162.72) | 485.31 (130.10) | 498.46 (142.04)
    Treatment-Naive Participants: number analyzed (Participants) | 58 | 54 | 51 | 163
    Treatment-Naive Participants | 490.88 (139.01) | 535.44 (163.13) | 496.47 (134.96) | 507.39 (146.71)
    Previously Treated Participants: number analyzed (Participants) | 31 | 1 | 29 | 61
    Previously Treated Participants | 485.52 (134.56) | 395.00 (NA) — Standard deviation could not be calculated from data for a single participant. | 465.69 (120.86) | 474.61 (126.79)
Number of Participants with Absence/Presence of Subretinal Fluid in the Study Eye at Baseline [Count of Participants; unit: Participants] — Subretinal fluid is defined as the presence of fluid between the retina and the retinal pigment epithelium. Resolution of subretinal fluid was measured using SD-OCT. Population: Baseline characteristics were analyzed for all participants, treatment-naive participants, and previously treated participants. This analysis included participants who had received at least one dose of study drug and had non-missing assessments at baseline.
  Participants
    All Participants: number analyzed (Participants) | 89 | 55 | 80 | 224
    All Participants: Subretinal Fluid Absent | 49 | 30 | 44 | 123
    All Participants: Subretinal Fluid Present | 40 | 25 | 36 | 101
    Treatment-Naive Participants: number analyzed (Participants) | 58 | 54 | 51 | 163
    Treatment-Naive Participants: Subretinal Fluid Absent | 34 | 30 | 25 | 89
    Treatment-Naive Participants: Subretinal Fluid Present | 24 | 24 | 26 | 74
    Previously Treated Participants: number analyzed (Participants) | 31 | 1 | 29 | 61
    Previously Treated Participants: Subretinal Fluid Absent | 15 | 0 | 19 | 34
    Previously Treated Participants: Subretinal Fluid Present | 16 | 1 | 10 | 27
Number of Participants with Absence/Presence of Intraretinal Fluid at Baseline [Count of Participants; unit: Participants] — Intraretinal fluid is described as the presence of fluid within the retina. Resolution of intraretinal fluid was measured by SD-OCT. Population: Baseline characteristics were analyzed for all participants, treatment-naive participants, and previously treated participants. This analysis included participants who had received at least one dose of study drug and had non-missing assessments at baseline.
  Participants
    All Participants: number analyzed (Participants) | 88 | 55 | 78 | 221
    All Participants: Intraretinal Fluid Absent | 1 | 0 | 0 | 1
    All Participants: Intraretinal Fluid Present | 87 | 55 | 78 | 220
    Treatment-Naive Participants: number analyzed (Participants) | 58 | 54 | 49 | 161
    Treatment-Naive Participants: Intraretinal Fluid Absent | 1 | 0 | 0 | 1
    Treatment-Naive Participants: Intraretinal Fluid Present | 57 | 54 | 49 | 160
    Previously Treated Participants: number analyzed (Participants) | 30 | 1 | 29 | 60
    Previously Treated Participants: Intraretinal Fluid Absent | 0 | 0 | 0 | 0
    Previously Treated Participants: Intraretinal Fluid Present | 30 | 1 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in BCVA Letter Score at Week 24, in Treatment-Naive Participants
Description: Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity examiner masked to study drug arm assignment. The BCVA examiner was masked to study eye and treatment assignment and only performed the refraction and BCVA assessment, but was not allowed to perform any other tasks involving direct care. The BCVA examiner was also masked to the BCVA letter scores of a participant's previous visits and could only know the participant's refraction data from previous visits. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The primary analysis used a Linear Mixed Effects Model for Repeated Measurements. Missing values were not imputed; it was assumed that the data were missing at random.
Time Frame: Baseline, Week 24
Population: Efficacy Population: all treatment-naive participants who had received at least one dose of study drug grouped by treatment assigned at randomization (did not differ from actual treatment during the study). This analysis only included participants with non-missing assessments at Baseline and Week 24.
Measure: Least Squares Mean (80% Confidence Interval); unit: BCVA letters
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 49 | 49 | 44
BCVA letters | 10.3 [8.8 to 11.9] | 11.7 [10.1 to 13.3] | 13.9 [12.2 to 15.6]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; Null hypothesis (H0): There is no difference between either of the faricimab treatment arms (Arms B and C) and the active comparator ranibizumab treatment arm (Arm A). The alternative hypothesis (Ha): Either of the faricimab treatment arms (Arm B or C) is different from the ranibizumab treatment arm (Arm A); Test type: Superiority; p = 0.37, Mixed Effects Model of Repeated Measures — There was no formal correction for multiple comparisons. Test for Arm B vs. Arm A was carried out at one-sided 10% alpha; Categorical covariates: treatment group, categorical visit, and visit by treatment group, stratification factors; continuous covariate: baseline BCVA; Difference in Least Squares Means = 1.4, 80% CI 2-sided [-0.6 to 3.4] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.03, Mixed Effects Model of Repeated Measures — There was no formal correction for multiple comparisons. Test for Arm C vs. Arm A was carried out at one-sided 10% alpha; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 3.6, 80% CI 2-sided [1.5 to 5.6] — The mean difference between arms was calculated as Arm C minus Arm A

2. Secondary Outcome: Mean Change From Baseline in BCVA Letter Score at Week 24, in Previously Treated Participants
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Efficacy Population: all previously treated participants who had received at least one dose of study drug grouped by treatment assigned at randomization (did not differ from actual treatment during the study). This analysis only included participants with non-missing assessments at Baseline and Week 24.
Measure: Least Squares Mean (80% Confidence Interval); unit: BCVA letters
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 28 | 23
BCVA letters | 8.9 [5.7 to 10.8] | 9.6 [7.0 to 12.3]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; Null hypothesis (H0): There is no difference between either of the faricimab treatment arm (Arm C) and the active comparator ranibizumab treatment arm (Arm A). The alternative hypothesis (Ha): The faricimab treatment arms (Arm C) is different from the ranibizumab treatment arm (Arm A); Test type: Superiority; p = 0.63, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 1.3, 80% CI 2-sided [-2.3 to 5.0] — The mean difference between arms was calculated as Arm C minus Arm A

3. Secondary Outcome: Mean Change From Baseline in BCVA Letter Score at Week 24, in All Participants
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Efficacy Population: all participants who had received at least one dose of study drug grouped by treatment assigned at randomization (did not differ from actual treatment during the study). This analysis only included participants with non-missing assessments at Baseline and Week 24.
Measure: Least Squares Mean (80% Confidence Interval); unit: BCVA letters
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 77 | 50 | 67
BCVA letters | 9.4 [8.1 to 10.7] | 11.7 [10.0 to 13.4] | 12.3 [10.9 to 13.7]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.15, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.3, 80% CI 2-sided [0.2 to 4.3] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.04, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.9, 80% CI 2-sided [1.1 to 4.7] — The mean difference between arms was calculated as Arm C minus Arm A

4. Secondary Outcome: Mean Percentage of Participants Who Gained ≥15 ETDRS Letters From Baseline BCVA Score at Week 24, in Treatment-Naive Participants
Description: Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity examiner masked to study drug arm assignment. The BCVA examiner was masked to study eye and treatment assignment and only performed the refraction and BCVA assessment, but was not allowed to perform any other tasks involving direct care. The BCVA examiner was also masked to the BCVA letter scores of a participant's previous visits and could only know the participant's refraction data from previous visits. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The outcome measure was analyzed using a Generalized Estimating Equations Model. Missing values were not imputed; it was assumed that the data were missing at random.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 49 | 49 | 44
Percentage of participants | 35.3 [27.3 to 44.1] | 36.0 [27.9 to 45.0] | 42.5 [33.5 to 52.1]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.94, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = 0.8, 80% CI 2-sided [-11.3 to 12.8] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.46, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 2]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = 7.3, 80% CI 2-sided [-5.4 to 19.9] — The mean difference between arms was calculated as Arm C minus Arm A

5. Secondary Outcome: Mean Percentage of Participants Who Gained ≥15 ETDRS Letters From Baseline BCVA Score at Week 24, in Previously Treated Participants
Description: as for outcome 4
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 28 | 23
Percentage of participants | 16.8 [9.6 to 27.8] | 23.2 [14.1 to 35.7]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.56, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 2]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Percentage of Participants = 6.4, 80% CI 2-sided [-7.7 to 20.5] — The mean difference between arms was calculated as Arm C minus Arm A

6. Secondary Outcome: Mean Percentage of Participants Who Gained ≥15 ETDRS Letters From Baseline BCVA Score at Week 24, in All Participants
Description: as for outcome 4
Time Frame: Baseline up to Week 24
Population: as for outcome 3
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 77 | 50 | 67
Percentage of participants | 28.7 [22.7 to 35.5] | 35.3 [27.4 to 44.2] | 35.9 [28.9 to 43.6]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.43, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = 6.6, 80% CI 2-sided [-4.0 to 17.2] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.34, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 2]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = 7.2, 80% CI 2-sided [-2.6 to 17.0] — The mean difference between arms was calculated as Arm C minus Arm A

7. Secondary Outcome: Mean Percentage of Participants With BCVA ≥69 Letters (20/40 or Better) at Week 24, in Treatment-Naive Participants
Description: as for outcome 4
Time Frame: Week 24
Population: Efficacy Population: all treatment-naive participants who had received at least one dose of study drug grouped by treatment assigned at randomization (did not differ from actual treatment during the study). This analysis only included participants with non-missing assessments at Week 24.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 49 | 49 | 44
Percentage of participants | 69.0 [60.2 to 76.7] | 78.5 [70.3 to 84.9] | 75.8 [66.8 to 83.0]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.27, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = 9.5, 80% CI 2-sided [-1.6 to 20.6] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.45, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 2]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = 6.8, 80% CI 2-sided [-4.9 to 18.5] — The mean difference between arms was calculated as Arm C minus Arm A

8. Secondary Outcome: Mean Percentage of Participants With BCVA ≥69 Letters (20/40 or Better) at Week 24, in Previously Treated Participants
Description: as for outcome 4
Time Frame: Week 24
Population: Efficacy Population: all previously treated participants who had received at least one dose of study drug grouped by treatment assigned at randomization (did not differ from actual treatment during the study). This analysis only included participants with non-missing assessments at Week 24.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 28 | 23
Percentage of participants | 69.0 [57.3 to 78.7] | 68.4 [55.4 to 79.0]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.96, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 2]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = -0.6, 80% CI 2-sided [-16.8 to 15.5] — The mean difference between arms was calculated as Arm C minus Arm A

9. Secondary Outcome: Mean Percentage of Participants With BCVA ≥69 Letters (20/40 or Better) at Week 24, in All Participants
Description: as for outcome 4
Time Frame: Week 24
Population: Efficacy Population: all participants who had received at least one dose of study drug grouped by treatment assigned at randomization (did not differ from actual treatment during the study). This analysis only included participants with non-missing assessments at Week 24.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 77 | 50 | 67
Percentage of participants | 69.0 [62.1 to 75.2] | 78.9 [70.8 to 85.2] | 73.2 [65.9 to 79.4]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.19, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = 9.9, 80% CI 2-sided [0.1 to 19.7] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.57, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 2]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = 4.2, 80% CI 2-sided [-5.3 to 13.6] — The mean difference between arms was calculated as Arm C minus Arm A

10. Secondary Outcome: Mean Percentage of Participants With BCVA ≥84 Letters (20/20 or Better) at Week 24, in Treatment-Naive Participants
Description: as for outcome 4
Time Frame: Week 24
Population: as for outcome 7
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 49 | 49 | 44
Percentage of participants | 11.5 [6.9 to 18.7] | 8.7 [4.8 to 15.3] | 9.8 [5.5 to 16.8]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.64, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = -2.8, 80% CI 2-sided [-10.5 to 4.9] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.78, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 2]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = -1.8, 80% CI 2-sided [-9.8 to 6.2] — The mean difference between arms was calculated as Arm C minus Arm A

11. Secondary Outcome: Mean Percentage of Participants With BCVA ≥84 Letters (20/20 or Better) at Week 24, in Previously Treated Participants
Description: as for outcome 4
Time Frame: Week 24
Population: as for outcome 8
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 28 | 23
Percentage of participants | 10.5 [5.0 to 20.6] | 8.2 [3.3 to 19.1]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.78, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 2]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = -2.3, 80% CI 2-sided [-12.7 to 8.2] — The mean difference between arms was calculated as Arm C minus Arm A

12. Secondary Outcome: Mean Percentage of Participants With BCVA ≥84 Letters (20/20 or Better) at Week 24, in All Participants
Description: as for outcome 4
Time Frame: Week 24
Population: as for outcome 9
Measure: Least Squares Mean (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 77 | 50 | 67
Percentage of participants | 11.1 [7.3 to 16.6] | 10.6 [6.2 to 17.5] | 9.1 [5.6 to 14.6]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.93, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 1]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = -0.5, 80% CI 2-sided [-7.7 to 6.7] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.69, Generalized Estimating Equations Model — [p-value comment as in outcome 1, analysis 2]; Categorical covariates: treatment group, visit, and visit by treatment group interaction term; Difference in Least Squares Means = -2.0, 80% CI 2-sided [-8.3 to 4.4] — The mean difference between arms was calculated as Arm C minus Arm A

13. Secondary Outcome: Mean Change From Baseline in Foveal Center Point Thickness at Week 24, in Treatment-Naive Participants
Description: Foveal center point thickness (FCPT) is defined as the thickness from the inner limiting membrane to the retinal pigment epithelial at the horizontal slice closest to the center of the fovea. Foveal center point thickness was measured using spectral domain optical coherence tomography (SD-OCT).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (80% Confidence Interval); unit: micrometers
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 49 | 49 | 44
micrometers | -243.4 [-261.2 to -225.2] | -249.9 [-269.5 to -230.4] | -266.2 [-286.6 to -245.8]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.69, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Categorical covariates: treatment group, categorical visit, and visit by treatment group, stratification factors; continuous covariate: baseline FCPT; Difference in Least Squares Means = -6.5, 80% CI 2-sided [-27.8 to 14.7] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.18, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 13, analysis 1]; Difference in Least Squares Means = -22.8, 80% CI 2-sided [-44.5 to -1.2] — The mean difference between arms was calculated as Arm C minus Arm A

14. Secondary Outcome: Mean Change From Baseline in Foveal Center Point Thickness at Week 24, in Previously Treated Participants
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: micrometers
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 28 | 23
micrometers | -162.1 [-186.9 to -137.3] | -211.3 [-237.1 to -185.5]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.07, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 13, analysis 1]; Difference in Least Squares Means = -49.2, 80% CI 2-sided [-84.2 to -14.2] — The mean difference between arms was calculated as Arm C minus Arm A

15. Secondary Outcome: Mean Change From Baseline in Foveal Center Point Thickness at Week 24, in All Participants
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (80% Confidence Interval); unit: micrometers
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 77 | 50 | 67
micrometers | -210.7 [-225.0 to -196.4] | -228.0 [-246.4 to -209.7] | -239.9 [-255.2 to -224.6]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.28, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 13, analysis 1]; Difference in Least Squares Means = -17.3, 80% CI 2-sided [-38.0 to 3.4] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 13, analysis 1]; Difference in Least Squares Means = -29.2, 80% CI 2-sided [-47.8 to -10.6] — The mean difference between arms was calculated as Arm C minus Arm A

16. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness at Week 24, in Treatment-Naive Participants
Description: Central subfield thickness (CST) is defined as the mean thickness from the inner limiting membrane to the retinal pigment epithelial over the 1 millimetre (mm) central subfield. Central subfield thickness was measured using SD-OCT.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (80% Confidence Interval); unit: micrometers
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 49 | 49 | 44
micrometers | -204.7 [-219.6 to -189.8] | -217.1 [-233.0 to -201.2] | -225.8 [-242.5 to -209.1]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.36, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Categorical covariates: treatment group, categorical visit, and visit by treatment group, stratification factors; continuous covariate: baseline CST; Difference in Least Squares Means = -12.4, 80% CI 2-sided [-29.7 to 5.0] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.13, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 16, analysis 1]; Difference in Least Squares Means = -21.1, 80% CI 2-sided [-38.7 to -3.5] — The mean difference between arms was calculated as Arm C minus Arm A

17. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness at Week 24, in Previously Treated Participants
Description: as for outcome 16
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: micrometers
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 28 | 23
micrometers | -148.0 [-167.7 to -128.4] | -186.6 [-206.9 to -166.4]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.07, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 16, analysis 1]; Difference in Least Squares Means = -38.6, 80% CI 2-sided [-65.9 to -11.3] — The mean difference between arms was calculated as Arm C minus Arm A

18. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness at Week 24, in All Participants
Description: as for outcome 16
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (80% Confidence Interval); unit: micrometers
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 77 | 50 | 67
micrometers | -180.2 [-191.6 to -168.8] | -200.3 [-214.8 to -185.8] | -206.9 [-219.0 to -194.8]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.12, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Difference in Least Squares Means = -20.1, 80% CI 2-sided [-36.4 to -3.8] — The mean difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.02, Mixed Effects Model of Repeated Measures — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 16, analysis 1]; Difference in Least Squares Means = -26.7, 80% CI 2-sided [-41.3 to -12.0] — The mean difference between arms was calculated as Arm C minus Arm A

19. Secondary Outcome: Percentage of Participants With Presence of Subretinal Fluid in the Study Eye at Week 24, in Treatment-Naive Participants
Description: Subretinal fluid is defined as the presence of fluid between the retina and the retinal pigment epithelium. Resolution of subretinal fluid was measured using SD-OCT.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 49 | 49 | 44
Percentage of participants | 4.08 [0.46 to 7.70] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4948, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = -4.08, 80% CI 2-sided [-7.70 to -0.46] — The difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4960, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Difference in Percentage of Participants = -4.08, 80% CI 2-sided [-7.70 to -0.46] — The difference between arms was calculated as Arm C minus Arm A

20. Secondary Outcome: Percentage of Participants With Presence of Subretinal Fluid in the Study Eye at Week 24, in Previously Treated Participants
Description: as for outcome 19
Time Frame: Week 24
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 28 | 23
Percentage of participants | 7.14 [0.91 to 13.38] | 4.35 [0.00 to 9.80]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 1.0000, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Difference in Percentage of Participants = -2.80, 80% CI 2-sided [-11.08 to 5.49] — The difference between arms was calculated as Arm C minus Arm A

21. Secondary Outcome: Percentage of Participants With Presence of Intraretinal Fluid in the Study Eye at Week 24, in Treatment-Naive Participants
Description: Intraretinal fluid is described as the presence of fluid within the retina. Resolution of intraretinal fluid was measured by SD-OCT.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 49 | 49 | 44
percentage of participants | 87.76 [81.75 to 93.76] | 81.63 [74.54 to 88.72] | 90.91 [85.35 to 96.46]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm B: 1.5 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5759, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = -6.12, 80% CI 2-sided [-15.41 to 3.17] — The difference between arms was calculated as Arm B minus Arm A
Statistical Analysis 2: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7437, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Difference in Percentage of Participants = 3.15, 80% CI 2-sided [-5.02 to 11.33] — The difference between arms was calculated as Arm C minus Arm A

22. Secondary Outcome: Percentage of Participants With Presence of Intraretinal Fluid in the Study Eye at Week 24, in Previously Treated Participants
Description: as for outcome 21
Time Frame: Week 24
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 28 | 23
percentage of participants | 89.29 [81.79 to 96.78] | 91.30 [83.77 to 98.83]
Statistical Analysis 1: Comparison: Arm A: 0.3 mg Ranibizumab vs Arm C: 6 mg Faricimab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 1.0000, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Difference in Percentage of Participants = 2.02, 80% CI 2-sided [-8.60 to 12.64] — The difference between arms was calculated as Arm C minus Arm A

23. Secondary Outcome: Number of Participants With Presence or Absence of Leakage at the Macula at Week 24, in Treatment-Naive Participants
Description: Leakage at the macula describes the leakage of fluorescein at the macula region as measured by fundus fluorescein angiography (FFA).
Time Frame: Week 24
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 45 | 46 | 36
Participants
  Leakage Present | 41 | 41 | 25
  Leakage Absent | 4 | 5 | 11

24. Secondary Outcome: Number of Participants With Presence or Absence of Leakage at the Macula at Week 24, in Previously Treated Participants
Description: as for outcome 23
Time Frame: Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 25 | 1 | 16
Participants
  Leakage Present | 24 | 1 | 14
  Leakage Absent | 1 | 0 | 2

25. Secondary Outcome: Mean Change From Baseline in the Size of the Foveal Avascular Zone at Week 24, in All Participants
Description: The size of the foveal avascular zone was to be measured by fundus fluorescein angiography (FFA).
Time Frame: Baseline, Week 24
Population: Due to the poor image quality available, size of the foveal avascular zone could not be assessed in any of the participant populations.
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Mean Plasma Concentrations of Ranibizumab (Arm A) or Faricimab (Arms B and C) Over Time, in All Participants
Description: Plasma concentrations of ranibizumab were measured by an appropriate assay only from samples of participants randomized to Arm A: 0.3 mg Ranibizumab. Plasma concentrations of faricimab were measured by a specific validated enzyme-linked immunoabsorbent assay (ELISA) only from samples of participants randomized to Arm B: 1.5 mg Faricimab and Arm C: 6 mg Faricimab. Baseline was defined as the last non-missing predose assessment. The lower limit of quantification (LLOQ) for the ranibizumab and faricimab assays were 0.015 nanograms per millilitre (ng/mL) and 0.800 ng/mL, respectively. Values below the limit of quantification were imputed as LLOQ divided by 2.
Time Frame: Predose at Baseline and Weeks 1, 4, 12, 20, 24, 26, 28, 32, and 36
Population: Pharmacokinetics Population: The analysis included participants who received at least one dose of study drug grouped by treatment assigned at randomization (did not differ from actual treatment during the study) and had plasma samples available at a given study visit timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 90 | 55 | 82
nanograms per millilitre (ng/mL)
  Baseline: number analyzed (Participants) | 34 | 54 | 78
  Baseline | 2.20 (7.84) | 0.40 (0.00) | 0.40 (0.00)
  Week 1: number analyzed (Participants) | 32 | 52 | 68
  Week 1 | 2.52 (7.57) | 48.36 (22.46) | 172.24 (80.59)
  Week 4: number analyzed (Participants) | 33 | 53 | 76
  Week 4 | 0.86 (2.27) | 6.97 (4.96) | 20.60 (13.46)
  Week 12: number analyzed (Participants) | 32 | 51 | 71
  Week 12 | 0.26 (0.48) | 9.32 (5.93) | 22.38 (13.63)
  Week 20: number analyzed (Participants) | 28 | 52 | 70
  Week 20 | 0.21 (0.35) | 7.11 (4.64) | 22.59 (18.10)
  Week 24: number analyzed (Participants) | 34 | 49 | 64
  Week 24 | 0.20 (0.44) | 8.69 (5.06) | 20.18 (16.37)
  Week 26: number analyzed (Participants) | 25 | 13 | 25
  Week 26 | 0.19 (0.47) | 3.80 (3.28) | 8.18 (6.98)
  Week 28: number analyzed (Participants) | 28 | 13 | 29
  Week 28 | 0.10 (0.16) | 1.44 (2.42) | 2.94 (3.07)
  Week 32: number analyzed (Participants) | 22 | 15 | 22
  Week 32 | 0.05 (0.09) | 0.46 (0.23) | 0.82 (0.97)
  Week 36: number analyzed (Participants) | 21 | 37 | 53
  Week 36 | 0.03 (0.05) | 0.40 (0.00) | 0.40 (0.00)

27. Secondary Outcome: Baseline and Change From Baseline in Free Vascular Endothelial Growth Factor (VEGF) Plasma Levels Over Time, in Treatment-Naive Participants
Description: The concentration of free VEGF was determined in plasma samples using an enzyme-linked immunosorbent assay (ELISA) method. The lower limit of quantification (LLOQ) of the assay was 15.6 picograms per millilitre (pg/mL). Plasma free VEGF concentrations below the limit of quantification were imputed as LLOQ divided by 2.
Time Frame: Baseline and Weeks 1, 4, 12, 16, 24, 26, 28, 32, and 36
Population: Pharmacodynamics Population: The analysis included participants who received at least one dose of study drug grouped by treatment assigned at randomization (did not differ from actual treatment during the study) and had plasma samples available at a given study visit timepoint.
Measure: Mean (Standard Deviation); unit: picograms per millilitre (pg/mL)
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 59 | 54 | 53
picograms per millilitre (pg/mL)
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 54 | 51 | 48
  Baseline (BL) - Value at Visit | 23.93 (52.75) | 14.93 (19.70) | 12.45 (7.62)
  Change from BL at Week 1: number analyzed (Participants) | 49 | 49 | 44
  Change from BL at Week 1 | -9.44 (49.77) | -3.85 (20.99) | -3.61 (6.96)
  Change from BL at Week 4: number analyzed (Participants) | 51 | 50 | 48
  Change from BL at Week 4 | -1.68 (21.20) | -0.37 (21.76) | -0.49 (9.31)
  Change from BL at Week 12: number analyzed (Participants) | 47 | 47 | 44
  Change from BL at Week 12 | -3.54 (22.50) | -1.61 (20.82) | 1.67 (16.69)
  Change from BL at Week 16: number analyzed (Participants) | 0 | 1 | 0
  Change from BL at Week 16 |  | 0.00 (NA) — Standard deviation could not be calculated using data from a single participant. |
  Change from BL at Week 24: number analyzed (Participants) | 43 | 43 | 41
  Change from BL at Week 24 | -7.31 (23.97) | 2.92 (18.23) | 2.83 (13.74)
  Change from BL at Week 26: number analyzed (Participants) | 15 | 12 | 15
  Change from BL at Week 26 | -4.37 (13.09) | -2.98 (6.27) | -2.43 (7.08)
  Change from BL at Week 28: number analyzed (Participants) | 6 | 7 | 4
  Change from BL at Week 28 | 0.30 (5.87) | 0.73 (12.17) | 7.15 (7.73)
  Change from BL at Week 32: number analyzed (Participants) | 4 | 4 | 4
  Change from BL at Week 32 | -3.30 (8.13) | -35.85 (65.08) | 4.50 (5.97)
  Change from BL at Week 36: number analyzed (Participants) | 30 | 34 | 33
  Change from BL at Week 36 | -1.75 (14.00) | 0.69 (7.71) | 2.07 (10.38)

28. Secondary Outcome: Baseline and Change From Baseline in Free Vascular Endothelial Growth Factor (VEGF) Plasma Levels Over Time, in Previously Treated Participants
Description: as for outcome 27
Time Frame: Baseline and Weeks 1, 4, 12, 16, 24, 26, 28, 32, and 36
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: picograms per millilitre (pg/mL)
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 31 | 1 | 29
picograms per millilitre (pg/mL)
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 28 | 1 | 26
  Baseline (BL) - Value at Visit | 12.94 (10.00) | 7.80 (NA) — Standard deviation could not be calculated using data from a single participant. | 16.21 (10.22)
  Change from BL at Week 1: number analyzed (Participants) | 26 | 1 | 22
  Change from BL at Week 1 | 0.50 (14.24) | 8.20 (NA) — Standard deviation could not be calculated using data from a single participant. | -7.40 (12.08)
  Change from BL at Week 4: number analyzed (Participants) | 28 | 1 | 26
  Change from BL at Week 4 | 0.93 (15.07) | 14.50 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.80 (11.11)
  Change from BL at Week 12: number analyzed (Participants) | 28 | 1 | 24
  Change from BL at Week 12 | 13.83 (51.87) | 39.20 (NA) — Standard deviation could not be calculated using data from a single participant. | 0.78 (16.55)
  Change from BL at Week 16: number analyzed (Participants) | 0 | 0 | 1
  Change from BL at Week 16 |  |  | 19.10 (NA) — Standard deviation could not be calculated using data from a single participant.
  Change from BL at Week 24: number analyzed (Participants) | 24 | 1 | 21
  Change from BL at Week 24 | 6.60 (31.50) | 12.40 (NA) — Standard deviation could not be calculated using data from a single participant. | 4.13 (27.51)
  Change from BL at Week 26: number analyzed (Participants) | 10 | 0 | 6
  Change from BL at Week 26 | -0.25 (13.97) |  | 16.65 (42.34)
  Change from BL at Week 28: number analyzed (Participants) | 6 | 0 | 2
  Change from BL at Week 28 | 7.32 (20.30) |  | 0.00 (0.00)
  Change from BL at Week 32: number analyzed (Participants) | 3 | 0 | 1
  Change from BL at Week 32 | -1.13 (11.24) |  | 57.00 (NA) — Standard deviation could not be calculated using data from a single participant.
  Change from BL at Week 36: number analyzed (Participants) | 18 | 1 | 18
  Change from BL at Week 36 | 3.05 (11.44) | 21.50 (NA) — Standard deviation could not be calculated using data from a single participant. | 3.53 (21.58)

29. Secondary Outcome: Baseline and Change From Baseline in Total Angiopoietin-2 (Ang-2) Plasma Levels Over Time, in Treatment-Naive Participants
Description: Total Ang-2 concentrations were determined in plasma samples using an appropriate assay method. The lower limit of quantification (LLOQ) of the assay was 0.09 nanograms per millilitre (ng/mL). Plasma total Ang-2 concentrations below the limit of quantification were imputed as LLOQ divided by 2.
Time Frame: Baseline and Weeks 1, 4, 12, 16, 24, 26, 28, 32, and 36
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 59 | 54 | 53
nanograms per millilitre (ng/mL)
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 53 | 51 | 49
  Baseline (BL) - Value at Visit | 2.77 (2.01) | 2.07 (0.91) | 2.30 (1.88)
  Change from BL at Week 1: number analyzed (Participants) | 48 | 48 | 45
  Change from BL at Week 1 | 0.07 (0.60) | 0.04 (0.80) | 0.75 (0.79)
  Change from BL at Week 4: number analyzed (Participants) | 50 | 49 | 48
  Change from BL at Week 4 | 0.14 (0.72) | 0.05 (0.63) | 0.24 (0.79)
  Change from BL at Week 12: number analyzed (Participants) | 47 | 48 | 46
  Change from BL at Week 12 | 0.06 (0.66) | 0.14 (0.51) | 0.18 (1.02)
  Change from BL at Week 16: number analyzed (Participants) | 0 | 1 | 0
  Change from BL at Week 16 |  | -0.08 (NA) — Standard deviation could not be calculated using data from a single participant. |
  Change from BL at Week 24: number analyzed (Participants) | 23 | 35 | 35
  Change from BL at Week 24 | 0.30 (0.80) | 0.40 (0.90) | 0.00 (0.61)
  Change from BL at Week 26: number analyzed (Participants) | 15 | 13 | 15
  Change from BL at Week 26 | 0.25 (1.37) | 0.21 (0.33) | 0.58 (0.78)
  Change from BL at Week 28: number analyzed (Participants) | 6 | 5 | 4
  Change from BL at Week 28 | 0.11 (0.35) | 0.34 (0.35) | -0.20 (0.49)
  Change from BL at Week 32: number analyzed (Participants) | 4 | 5 | 4
  Change from BL at Week 32 | -0.35 (0.50) | 1.58 (1.91) | 0.42 (0.21)
  Change from BL at Week 36: number analyzed (Participants) | 29 | 34 | 34
  Change from BL at Week 36 | 0.05 (0.83) | 0.39 (1.45) | -0.02 (0.83)

30. Secondary Outcome: Baseline and Change From Baseline in Free Angiopoietin-2 (Ang-2) Plasma Levels Over Time, in Treatment-Naive Participants
Description: Free Ang-2 concentrations were determined in plasma samples using an appropriate assay method. The lower limit of quantification (LLOQ) of the assay was 0.9 nanograms per millilitre (ng/mL). Plasma free Ang-2 concentrations below the limit of quantification were imputed as LLOQ divided by 2.
Time Frame: Baseline and Weeks 1, 4, 12, 16, 24, 26, 28, 32, and 36
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 59 | 54 | 53
nanograms per millilitre (ng/mL)
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 53 | 51 | 49
  Baseline (BL) - Value at Visit | 3.05 (1.72) | 2.38 (1.04) | 2.46 (1.37)
  Change from BL at Week 1: number analyzed (Participants) | 48 | 48 | 45
  Change from BL at Week 1 | -0.49 (0.46) | -0.59 (0.79) | 0.06 (1.01)
  Change from BL at Week 4: number analyzed (Participants) | 50 | 49 | 48
  Change from BL at Week 4 | -0.36 (0.66) | -0.45 (0.72) | -0.22 (0.88)
  Change from BL at Week 12: number analyzed (Participants) | 47 | 48 | 46
  Change from BL at Week 12 | -0.07 (0.87) | 0.10 (0.68) | 0.25 (1.11)
  Change from BL at Week 16: number analyzed (Participants) | 0 | 1 | 0
  Change from BL at Week 16 |  | -0.74 (NA) — Standard deviation could not be calculated using data from a single participant. |
  Change from BL at Week 24: number analyzed (Participants) | 24 | 34 | 35
  Change from BL at Week 24 | -0.08 (0.95) | 0.19 (1.14) | -0.11 (0.86)
  Change from BL at Week 26: number analyzed (Participants) | 15 | 13 | 15
  Change from BL at Week 26 | -0.23 (1.27) | -0.26 (0.39) | 0.08 (0.76)
  Change from BL at Week 28: number analyzed (Participants) | 6 | 5 | 4
  Change from BL at Week 28 | -0.56 (0.69) | -0.37 (0.44) | -0.54 (0.60)
  Change from BL at Week 32: number analyzed (Participants) | 4 | 5 | 4
  Change from BL at Week 32 | -0.61 (0.58) | 0.92 (1.83) | -0.12 (0.28)
  Change from BL at Week 36: number analyzed (Participants) | 29 | 34 | 34
  Change from BL at Week 36 | -0.61 (0.87) | -0.15 (1.03) | -0.26 (0.89)

31. Secondary Outcome: Baseline and Change From Baseline in Total Angiopoietin-2 (Ang-2) Plasma Levels Over Time, in Previously Treated Participants
Description: as for outcome 29
Time Frame: Baseline and Weeks 1, 4, 12, 16, 24, 26, 28, 32, and 36
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 31 | 1 | 29
nanograms per millilitre (ng/mL)
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 29 | 1 | 26
  Baseline (BL) - Value at Visit | 2.40 (2.34) | 1.84 (NA) — Standard deviation could not be calculated using data from a single participant. | 2.31 (1.78)
  Change from BL at Week 1: number analyzed (Participants) | 26 | 1 | 21
  Change from BL at Week 1 | 0.15 (14.24) | 0.11 (NA) — Standard deviation could not be calculated using data from a single participant. | 0.94 (1.12)
  Change from BL at Week 4: number analyzed (Participants) | 28 | 1 | 26
  Change from BL at Week 4 | 0.03 (0.52) | -0.27 (NA) — Standard deviation could not be calculated using data from a single participant. | 0.14 (0.87)
  Change from BL at Week 12: number analyzed (Participants) | 28 | 1 | 24
  Change from BL at Week 12 | 0.33 (1.66) | -0.28 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.09 (0.46)
  Change from BL at Week 16: number analyzed (Participants) | 0 | 0 | 1
  Change from BL at Week 16 |  |  | -0.21 (NA) — Standard deviation could not be calculated using data from a single participant.
  Change from BL at Week 24: number analyzed (Participants) | 23 | 1 | 20
  Change from BL at Week 24 | 0.19 (1.22) | -0.19 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.16 (0.46)
  Change from BL at Week 26: number analyzed (Participants) | 10 | 0 | 6
  Change from BL at Week 26 | -0.07 (0.64) |  | -0.20 (0.42)
  Change from BL at Week 28: number analyzed (Participants) | 6 | 0 | 2
  Change from BL at Week 28 | 0.74 (2.78) |  | -0.91 (0.35)
  Change from BL at Week 32: number analyzed (Participants) | 4 | 0 | 1
  Change from BL at Week 32 | -0.04 (0.79) |  | 0.49 (NA) — Standard deviation could not be calculated using data from a single participant.
  Change from BL at Week 36: number analyzed (Participants) | 18 | 1 | 18
  Change from BL at Week 36 | 0.01 (0.72) | -0.47 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.13 (0.42)

32. Secondary Outcome: Baseline and Change From Baseline in Free Angiopoietin-2 (Ang-2) Plasma Levels Over Time, in Previously Treated Participants
Description: as for outcome 30
Time Frame: Baseline and Weeks 1, 4, 12, 16, 24, 26, 28, 32, and 36
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 31 | 1 | 29
nanograms per millilitre (ng/mL)
  Baseline (BL) - Value at Visit: number analyzed (Participants) | 29 | 1 | 27
  Baseline (BL) - Value at Visit | 2.67 (2.60) | 2.08 (NA) — Standard deviation could not be calculated using data from a single participant. | 2.35 (1.76)
  Change from BL at Week 1: number analyzed (Participants) | 26 | 1 | 22
  Change from BL at Week 1 | -0.07 (0.88) | -0.04 (NA) — Standard deviation could not be calculated using data from a single participant. | 0.30 (0.87)
  Change from BL at Week 4: number analyzed (Participants) | 28 | 1 | 27
  Change from BL at Week 4 | -0.33 (0.58) | -0.28 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.17 (0.66)
  Change from BL at Week 12: number analyzed (Participants) | 28 | 1 | 24
  Change from BL at Week 12 | -0.05 (1.12) | -0.65 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.13 (0.61)
  Change from BL at Week 16: number analyzed (Participants) | 0 | 0 | 1
  Change from BL at Week 16 |  |  | -0.49 (NA) — Standard deviation could not be calculated using data from a single participant.
  Change from BL at Week 24: number analyzed (Participants) | 21 | 1 | 19
  Change from BL at Week 24 | -0.28 (0.58) | -0.49 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.29 (0.64)
  Change from BL at Week 26: number analyzed (Participants) | 10 | 0 | 6
  Change from BL at Week 26 | -0.21 (0.79) |  | -0.16 (0.54)
  Change from BL at Week 28: number analyzed (Participants) | 6 | 0 | 2
  Change from BL at Week 28 | -0.17 (1.59) |  | -1.36 (0.83)
  Change from BL at Week 32: number analyzed (Participants) | 4 | 0 | 1
  Change from BL at Week 32 | -0.59 (0.68) |  | 0.07 (NA) — Standard deviation could not be calculated using data from a single participant.
  Change from BL at Week 36: number analyzed (Participants) | 18 | 1 | 18
  Change from BL at Week 36 | -0.29 (0.72) | -0.72 (NA) — Standard deviation could not be calculated using data from a single participant. | -0.19 (0.45)

33. Secondary Outcome: Safety Summary of the Number of Participants With at Least One Adverse Event During the Treatment Period (up to Week 24), in All Participants
Description: This safety summary reports the number and percentage of participants who experienced at least one adverse event (AE) within 28 days of the end of the treatment period (i.e., up to Week 24). AEs are categorized as any AEs, ocular AEs occurring in the study eye or fellow eye, systemic AEs, serious AEs, AEs related to treatment with study drug, AEs leading to discontinuation of treatment with study drug, and AEs with fatal outcome. Multiple occurrences of the same AE in one individual were counted only once.
Time Frame: From Baseline up to Week 24
Population: Safety Population: all participants who had received at least one dose of the study drug, whether prematurely withdrawn from the study or not, grouped according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  Any AE | 61 | 38 | 54
  Ocular AE | 30 | 21 | 32
  Ocular AE in the Study Eye | 22 | 16 | 22
  Related Ocular AE in the Study Eye | 1 | 0 | 2
  Ocular AE in Study Eye Leading to Discontinuation | 1 | 0 | 0
  Serious Ocular AE in the Study Eye | 1 | 0 | 1
  Ocular AE in the Fellow Eye | 19 | 14 | 18
  Systemic AE | 51 | 30 | 46
  Related Systemic AE | 0 | 0 | 2
  Serious Systemic AE | 8 | 6 | 7
  Systemic AE Leading to Discontinuation | 0 | 1 | 0
  Any Related AE | 1 | 0 | 4
  Any Serious AE | 9 | 7 | 8
  Any Related Serious AE | 0 | 0 | 0
  AE with Fatal Outcome | 2 | 1 | 2

34. Secondary Outcome: Safety Summary of the Number of Participants With at Least One Adverse Event During the Post-Treatment Observation Period, in All Participants
Description: This safety summary reports the number and percentage of participants who experienced at least one adverse event (AE) during the post-treatment observation period (i.e., from Week 24 up to Week 36). AEs are categorized as any AEs, ocular AEs occurring in the study eye or fellow eye, systemic AEs, serious AEs, AEs related to treatment with study drug, AEs leading to discontinuation of treatment with study drug, and AEs with fatal outcome. Multiple occurrences of the same AE in one individual were counted only once.
Time Frame: From Week 24 up to Week 36
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  Any AE | 31 | 21 | 34
  Ocular AE | 11 | 7 | 12
  Ocular AE in the Study Eye | 9 | 4 | 8
  Related Ocular AE in the Study Eye | 1 | 0 | 0
  Ocular AE in Study Eye Leading to Discontinuation | 0 | 0 | 0
  Serious Ocular AE in the Study Eye | 0 | 0 | 1
  Ocular AE in the Fellow Eye | 6 | 5 | 8
  Systemic AE | 22 | 15 | 25
  Related Systemic AE | 0 | 0 | 0
  Serious Systemic AE | 2 | 3 | 4
  Systemic AE Leading to Discontinuation | 0 | 0 | 0
  Any Related AE | 1 | 0 | 0
  Any Serious AE | 2 | 3 | 5
  Any Related Serious AE | 0 | 0 | 0
  AE with Fatal Outcome | 0 | 0 | 0

35. Secondary Outcome: Number of Participants With at Least One Ocular Adverse Event in the Study Eye or the Fellow Eye During the Treatment Period by Highest Intensity, in All Participants
Description: The investigator assessed adverse event severity according to the following grading scale: Mild = Discomfort noticed, but no disruption of normal daily activity; Moderate = Discomfort sufficient to reduce or affect normal daily activity; Severe = Incapacitating with inability to work or to perform normal daily activity. Only the most severe intensity was counted for multiple occurrences of the same adverse event per participant at the preferred term level. Severity and seriousness are not synonymous; regardless of severity, some adverse events may have also met seriousness criteria.
Time Frame: From Baseline up to Week 24
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  Study Eye - Ocular AE of Any Intensity | 22 | 16 | 22
  Study Eye - Mild Ocluar AE | 20 | 15 | 21
  Study Eye - Moderate Ocular AE | 2 | 3 | 3
  Study Eye - Severe Ocular AE | 1 | 0 | 0
  Fellow Eye - Ocular AE of Any Intensity | 19 | 14 | 18
  Fellow Eye - Mild Ocular AE | 13 | 13 | 14
  Fellow Eye - Moderate Ocular AE | 7 | 1 | 5
  Fellow Eye - Severe Ocular AE | 0 | 1 | 0

36. Secondary Outcome: Number of Participants With at Least One Systemic Adverse Event During the Treatment Period by Highest Intensity, in All Participants
Description: as for outcome 35
Time Frame: From Baseline up to Week 24
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  Systemic AE of Any Intensity | 51 | 30 | 46
  Mild Systemic AE | 34 | 19 | 34
  Moderate Systemic AE | 26 | 18 | 22
  Severe Systemic AE | 9 | 4 | 5

37. Secondary Outcome: Number of Participants With Abnormal Systolic Blood Pressure Over Time, in All Participants
Description: Abnormal systolic blood pressure (supine) was defined as any value outside of the standard reference range, from <70 (low) to >180 (high) millimetres of mercury (mmHg) or a change from baseline of greater than 30 mmHg (decrease or increase). Baseline was defined as the last non-missing predose assessment. Not every abnormal vital sign qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 26, 28, 32, and 36
Population: Safety Population; the number of participants with an abnormal vital sign (numerator) is reported among the number analyzed (denominator), which represents the number of participants without the abnormal vital sign at baseline and who were evaluable at a given assessment timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  Week 1 - Low: number analyzed (Participants) | 82 | 53 | 71
  Week 1 - Low | 0 | 0 | 0
  Week 1 - High: number analyzed (Participants) | 82 | 53 | 70
  Week 1 - High | 1 | 3 | 0
  Week 4 - Low: number analyzed (Participants) | 87 | 55 | 80
  Week 4 - Low | 0 | 0 | 0
  Week 4 - High: number analyzed (Participants) | 87 | 55 | 78
  Week 4 - High | 0 | 0 | 1
  Week 8 - Low: number analyzed (Participants) | 86 | 55 | 76
  Week 8 - Low | 0 | 0 | 0
  Week 8 - High: number analyzed (Participants) | 86 | 55 | 75
  Week 8 - High | 1 | 0 | 2
  Week 12 - Low: number analyzed (Participants) | 84 | 53 | 75
  Week 12 - Low | 0 | 0 | 0
  Week 12 - High: number analyzed (Participants) | 84 | 53 | 74
  Week 12 - High | 1 | 0 | 2
  Week 16 - Low: number analyzed (Participants) | 83 | 53 | 75
  Week 16 - Low | 0 | 0 | 0
  Week 16 - High: number analyzed (Participants) | 83 | 53 | 74
  Week 16 - High | 0 | 1 | 1
  Week 20 - Low: number analyzed (Participants) | 80 | 53 | 73
  Week 20 - Low | 0 | 0 | 0
  Week 20 - High: number analyzed (Participants) | 80 | 53 | 72
  Week 20 - High | 3 | 2 | 3
  Week 24 - Low: number analyzed (Participants) | 77 | 50 | 67
  Week 24 - Low | 0 | 0 | 0
  Week 24 - High: number analyzed (Participants) | 77 | 50 | 66
  Week 24 - High | 2 | 2 | 2
  Week 26 - Low: number analyzed (Participants) | 30 | 14 | 28
  Week 26 - Low | 0 | 0 | 0
  Week 26 - High: number analyzed (Participants) | 30 | 14 | 27
  Week 26 - High | 0 | 0 | 0
  Week 28 - Low: number analyzed (Participants) | 76 | 49 | 67
  Week 28 - Low | 0 | 0 | 0
  Week 28 - High: number analyzed (Participants) | 76 | 49 | 66
  Week 28 - High | 1 | 1 | 1
  Week 32 - Low: number analyzed (Participants) | 60 | 44 | 65
  Week 32 - Low | 0 | 0 | 0
  Week 32 - High: number analyzed (Participants) | 60 | 44 | 64
  Week 32 - High | 4 | 1 | 2
  Week 36 - Low: number analyzed (Participants) | 53 | 39 | 57
  Week 36 - Low | 0 | 0 | 0
  Week 36 - High: number analyzed (Participants) | 53 | 39 | 56
  Week 36 - High | 1 | 0 | 2

38. Secondary Outcome: Number of Participants With Abnormal Diastolic Blood Pressure Over Time, in All Participants
Description: Abnormal diastolic blood pressure (supine) was defined as any value outside of the standard reference range, from <40 (low) to >110 (high) millimetres of mercury (mmHg) or a change from baseline of greater than 20 mmHg (decrease or increase). Baseline was defined as the last non-missing predose assessment. Not every abnormal vital sign qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 26, 28, 32, and 36
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  Week 1 - Low: number analyzed (Participants) | 82 | 53 | 71
  Week 1 - Low | 0 | 0 | 0
  Week 1 - High: number analyzed (Participants) | 82 | 53 | 71
  Week 1 - High | 1 | 0 | 0
  Week 4 - Low: number analyzed (Participants) | 87 | 55 | 80
  Week 4 - Low | 0 | 0 | 0
  Week 4 - High: number analyzed (Participants) | 87 | 55 | 79
  Week 4 - High | 0 | 0 | 0
  Week 8 - Low: number analyzed (Participants) | 86 | 55 | 76
  Week 8 - Low | 0 | 0 | 0
  Week 8 - High: number analyzed (Participants) | 86 | 55 | 75
  Week 8 - High | 0 | 0 | 0
  Week 12 - Low: number analyzed (Participants) | 84 | 53 | 75
  Week 12 - Low | 0 | 0 | 0
  Week 12 - High: number analyzed (Participants) | 84 | 53 | 74
  Week 12 - High | 0 | 0 | 2
  Week 16 - Low: number analyzed (Participants) | 83 | 53 | 75
  Week 16 - Low | 0 | 0 | 0
  Week 16 - High: number analyzed (Participants) | 83 | 53 | 74
  Week 16 - High | 0 | 0 | 0
  Week 20 - Low: number analyzed (Participants) | 80 | 53 | 73
  Week 20 - Low | 0 | 0 | 0
  Week 20 - High: number analyzed (Participants) | 80 | 53 | 72
  Week 20 - High | 1 | 0 | 1
  Week 24 - Low: number analyzed (Participants) | 77 | 50 | 67
  Week 24 - Low | 0 | 0 | 0
  Week 24 - High: number analyzed (Participants) | 77 | 50 | 66
  Week 24 - High | 1 | 0 | 0
  Week 26 - Low: number analyzed (Participants) | 30 | 14 | 28
  Week 26 - Low | 0 | 0 | 0
  Week 26 - High: number analyzed (Participants) | 30 | 14 | 27
  Week 26 - High | 1 | 0 | 0
  Week 28 - Low: number analyzed (Participants) | 76 | 49 | 67
  Week 28 - Low | 0 | 0 | 0
  Week 28 - High: number analyzed (Participants) | 76 | 49 | 66
  Week 28 - High | 0 | 0 | 0
  Week 32 - Low: number analyzed (Participants) | 60 | 44 | 65
  Week 32 - Low | 0 | 0 | 0
  Week 32 - High: number analyzed (Participants) | 60 | 44 | 64
  Week 32 - High | 1 | 1 | 0
  Week 36 - Low: number analyzed (Participants) | 53 | 39 | 57
  Week 36 - Low | 0 | 0 | 0
  Week 36 - High: number analyzed (Participants) | 53 | 39 | 56
  Week 36 - High | 0 | 0 | 1

39. Secondary Outcome: Number of Participants With an Abnormal Heart Rate Over Time, in All Participants
Description: Abnormal heart rate (supine) was defined as any value outside of the standard reference range, from <40 (low) to >100 (high) beats per minute. Baseline was defined as the last non-missing predose assessment. Not every abnormal vital sign qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 26, 28, 32, and 36
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  Week 1 - Low: number analyzed (Participants) | 82 | 53 | 71
  Week 1 - Low | 0 | 0 | 0
  Week 1 - High: number analyzed (Participants) | 81 | 53 | 69
  Week 1 - High | 0 | 0 | 1
  Week 4 - Low: number analyzed (Participants) | 87 | 55 | 80
  Week 4 - Low | 0 | 0 | 0
  Week 4 - High: number analyzed (Participants) | 86 | 55 | 78
  Week 4 - High | 1 | 0 | 0
  Week 8 - Low: number analyzed (Participants) | 86 | 55 | 76
  Week 8 - Low | 0 | 0 | 0
  Week 8 - High: number analyzed (Participants) | 85 | 55 | 74
  Week 8 - High | 0 | 0 | 0
  Week 12 - Low: number analyzed (Participants) | 84 | 53 | 75
  Week 12 - Low | 0 | 0 | 0
  Week 12 - High: number analyzed (Participants) | 83 | 53 | 73
  Week 12 - High | 1 | 0 | 1
  Week 16 - Low: number analyzed (Participants) | 83 | 53 | 75
  Week 16 - Low | 0 | 0 | 0
  Week 16 - High: number analyzed (Participants) | 82 | 53 | 73
  Week 16 - High | 2 | 0 | 3
  Week 20 - Low: number analyzed (Participants) | 80 | 53 | 73
  Week 20 - Low | 0 | 0 | 0
  Week 20 - High: number analyzed (Participants) | 80 | 53 | 71
  Week 20 - High | 1 | 0 | 1
  Week 24 - Low: number analyzed (Participants) | 77 | 50 | 67
  Week 24 - Low | 0 | 0 | 0
  Week 24 - High: number analyzed (Participants) | 77 | 50 | 65
  Week 24 - High | 1 | 0 | 2
  Week 26 - Low: number analyzed (Participants) | 30 | 14 | 28
  Week 26 - Low | 0 | 0 | 0
  Week 26 - High: number analyzed (Participants) | 30 | 14 | 28
  Week 26 - High | 2 | 0 | 1
  Week 28 - Low: number analyzed (Participants) | 76 | 49 | 67
  Week 28 - Low | 0 | 0 | 0
  Week 28 - High: number analyzed (Participants) | 76 | 49 | 65
  Week 28 - High | 0 | 0 | 2
  Week 32 - Low: number analyzed (Participants) | 60 | 44 | 65
  Week 32 - Low | 0 | 0 | 0
  Week 32 - High: number analyzed (Participants) | 60 | 44 | 63
  Week 32 - High | 1 | 0 | 0
  Week 36 - Low: number analyzed (Participants) | 53 | 39 | 57
  Week 36 - Low | 0 | 0 | 0
  Week 36 - High: number analyzed (Participants) | 53 | 39 | 55
  Week 36 - High | 0 | 0 | 0

40. Secondary Outcome: Number of Participants With Abnormal Body Temperature Over Time, in All Participants
Description: Abnormal body temperature (supine) was defined as any value outside of the standard reference range, from <36.5 (low) to >37.5 (high) degrees Celsius. Baseline was defined as the last non-missing predose assessment. Not every abnormal vital sign qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 26, 28, 32, and 36
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  Week 1 - Low: number analyzed (Participants) | 53 | 35 | 45
  Week 1 - Low | 8 | 4 | 7
  Week 1 - High: number analyzed (Participants) | 81 | 52 | 71
  Week 1 - High | 0 | 0 | 1
  Week 4 - Low: number analyzed (Participants) | 58 | 36 | 49
  Week 4 - Low | 13 | 2 | 8
  Week 4 - High: number analyzed (Participants) | 87 | 54 | 80
  Week 4 - High | 0 | 1 | 0
  Week 8 - Low: number analyzed (Participants) | 57 | 36 | 47
  Week 8 - Low | 14 | 4 | 9
  Week 8 - High: number analyzed (Participants) | 86 | 54 | 76
  Week 8 - High | 1 | 1 | 1
  Week 12 - Low: number analyzed (Participants) | 57 | 34 | 47
  Week 12 - Low | 9 | 4 | 14
  Week 12 - High: number analyzed (Participants) | 84 | 52 | 75
  Week 12 - High | 1 | 1 | 0
  Week 16 - Low: number analyzed (Participants) | 55 | 34 | 47
  Week 16 - Low | 5 | 3 | 13
  Week 16 - High: number analyzed (Participants) | 83 | 52 | 75
  Week 16 - High | 1 | 1 | 0
  Week 20 - Low: number analyzed (Participants) | 52 | 34 | 46
  Week 20 - Low | 8 | 6 | 7
  Week 20 - High: number analyzed (Participants) | 80 | 52 | 73
  Week 20 - High | 0 | 0 | 0
  Week 24 - Low: number analyzed (Participants) | 50 | 33 | 40
  Week 24 - Low | 13 | 6 | 10
  Week 24 - High: number analyzed (Participants) | 77 | 49 | 67
  Week 24 - High | 0 | 0 | 1
  Week 26 - Low: number analyzed (Participants) | 20 | 10 | 19
  Week 26 - Low | 3 | 1 | 5
  Week 26 - High: number analyzed (Participants) | 30 | 14 | 28
  Week 26 - High | 1 | 0 | 1
  Week 28 - Low: number analyzed (Participants) | 50 | 33 | 42
  Week 28 - Low | 11 | 4 | 10
  Week 28 - High: number analyzed (Participants) | 76 | 48 | 67
  Week 28 - High | 0 | 0 | 1
  Week 32 - Low: number analyzed (Participants) | 41 | 29 | 40
  Week 32 - Low | 7 | 7 | 9
  Week 32 - High: number analyzed (Participants) | 60 | 43 | 65
  Week 32 - High | 1 | 0 | 0
  Week 36 - Low: number analyzed (Participants) | 36 | 27 | 36
  Week 36 - Low | 5 | 7 | 8
  Week 36 - High: number analyzed (Participants) | 53 | 38 | 56
  Week 36 - High | 0 | 0 | 0

41. Secondary Outcome: Mean Heart Rate at Baseline and Week 24, as Measured by Electrocardiogram in All Participants
Description: Triplicate 12-lead electrocardiogram (ECG), i.e., three useful ECGs without artifacts, were performed on all evaluable participants. To minimize variability, it was important that participants be in a resting position for at least 10 minutes prior to the ECG evaluation. Body position was to be consistently maintained for each ECG evaluation to prevent changes in heart rate. Environmental distractions (e.g., television, radio, conversation, mobile phones) were to be minimized before and during ECG recording. Triplicate ECGs were to be obtained within a 5-minute interval. The predefined standard reference range for heart rate measured by ECG was 40 (low) to 100 (high) beats per minute.
Time Frame: Baseline, Week 24
Population: Safety Population: all participants who had received at least one dose of the study drug, whether prematurely withdrawn from the study or not, grouped according to the actual treatment received. This analysis included participants with non-missing assessments at Baseline and Week 24.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
beats per minute
  Baseline: number analyzed (Participants) | 87 | 54 | 78
  Baseline | 71.52 (14.47) | 73.65 (10.43) | 74.12 (12.89)
  Week 24: number analyzed (Participants) | 68 | 47 | 62
  Week 24 | 71.12 (12.53) | 73.96 (11.32) | 75.61 (11.46)

42. Secondary Outcome: Mean PR, RR, QT, QRS, QTcB, and QTcF Intervals at Baseline and Week 24, as Measured by Electrocardiogram in All Participants
Description: Triplicate 12-lead electrocardiogram (ECG), i.e., three useful ECGs without artifacts, were performed on all evaluable participants. To minimize variability, it was important that participants be in a resting position for at least 10 minutes prior to the ECG evaluation. Body position was to be consistently maintained for each ECG evaluation to prevent changes in heart rate. Environmental distractions (e.g., television, radio, conversation, mobile phones) were to be minimized before and during ECG recording. Triplicate ECGs were to be obtained within a 5-minute interval. Baseline was defined as the last non-missing predose assessment. The predefined standard reference ranges for the intervals measured by ECG were defined as follows (ranges are from low to high, in milliseconds [msec]): PR: 120-200 msec; RR: 600-1500 msec; QT: 200-500 msec; QRS: 40-120 msec.
Time Frame: Baseline, Week 24
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
milliseconds
  PR Interval at Baseline: number analyzed (Participants) | 82 | 54 | 75
  PR Interval at Baseline | 172.57 (28.62) | 168.50 (31.82) | 170.91 (29.06)
  PR Interval at Week 24: number analyzed (Participants) | 65 | 47 | 62
  PR Interval at Week 24 | 171.95 (30.21) | 167.49 (26.20) | 172.02 (28.81)
  RR Interval at Baseline: number analyzed (Participants) | 87 | 54 | 78
  RR Interval at Baseline | 864.44 (160.30) | 826.04 (119.67) | 828.64 (146.42)
  RR Interval at Week 24: number analyzed (Participants) | 68 | 47 | 62
  RR Interval at Week 24 | 864.34 (154.93) | 824.13 (126.72) | 806.45 (124.82)
  QT Interval at Baseline: number analyzed (Participants) | 87 | 54 | 78
  QT Interval at Baseline | 395.40 (40.47) | 387.87 (30.52) | 386.97 (32.65)
  QT Interval at Week 24: number analyzed (Participants) | 68 | 47 | 62
  QT Interval at Week 24 | 393.96 (36.74) | 384.30 (28.03) | 381.50 (28.10)
  QRS Interval at Baseline: number analyzed (Participants) | 87 | 54 | 78
  QRS Interval at Baseline | 98.84 (19.80) | 96.06 (16.76) | 95.26 (15.54)
  QRS Interval at Week 24: number analyzed (Participants) | 68 | 47 | 62
  QRS Interval at Week 24 | 98.82 (19.90) | 96.66 (11.24) | 95.40 (17.83)
  QTcB Interval at Baseline: number analyzed (Participants) | 87 | 54 | 78
  QTcB Interval at Baseline | 426.98 (24.47) | 427.85 (24.33) | 426.91 (22.84)
  QTcB Interval at Week 24: number analyzed (Participants) | 68 | 47 | 62
  QTcB Interval at Week 24 | 425.60 (25.55) | 424.79 (22.93) | 426.31 (23.36)
  QTcF Interval at Baseline: number analyzed (Participants) | 87 | 54 | 78
  QTcF Interval at Baseline | 415.60 (25.63) | 413.61 (23.15) | 412.67 (21.17)
  QTcF Interval at Week 24: number analyzed (Participants) | 68 | 47 | 62
  QTcF Interval at Week 24 | 414.21 (24.75) | 410.45 (20.35) | 410.42 (20.61)

43. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Hematology Tests, in All Participants
Description: Clinical laboratory tests for hematology parameters were performed and any marked abnormal values (High or Low) were based on Roche's predefined standard reference ranges. Marked laboratory abnormalities are presented according to COG3007 abnormality criteria: Single, Not Last = abnormality detected at a single assessment, but not at the last assessment; Last or Replicated = abnormality detected at the last assessment or replicated at one or more assessments. Not every laboratory abnormality qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy. Abs. = absolute count; Ery. = erythrocyte; Hemo. = hemoglobin
Time Frame: Predose at Baseline, Weeks 12 and 24, and at Early Termination and Unscheduled Visits (up to 36 weeks)
Population: Safety Population: all participants who had received at least one dose of the study drug, whether prematurely withdrawn from the study or not, grouped according to the actual treatment received. This analysis included participants with non-missing assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  Eosinophils, Abs., High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  Eosinophils, Abs., High - Any Abnormality | 2 | 1 | 3
  Eosinophils, Abs., High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  Eosinophils, Abs., High - Single, Not Last | 1 | 1 | 3
  Eosinophils, Abs., High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 72
  Eosinophils, Abs., High - Last or Replicated | 1 | 0 | 0
  Hematocrit, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  Hematocrit, Low - Any Abnormality | 4 | 1 | 1
  Hematocrit, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  Hematocrit, Low - Single, Not Last | 1 | 0 | 1
  Hematocrit, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 72
  Hematocrit, Low - Last or Replicated | 3 | 1 | 0
  Hemoglobin, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  Hemoglobin, Low - Any Abnormality | 4 | 1 | 2
  Hemoglobin, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  Hemoglobin, Low - Single, Not Last | 1 | 0 | 2
  Hemoglobin, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 72
  Hemoglobin, Low - Last or Replicated | 3 | 1 | 0
  Lymphocytes, Abs., Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  Lymphocytes, Abs., Low - Any Abnormality | 1 | 0 | 1
  Lymphocytes, Abs., Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  Lymphocytes, Abs., Low - Single, Not Last | 1 | 0 | 1
  Lymphocytes, Abs., Low - Last or Replicated: number analyzed (Participants) | 80 | 52 | 73
  Lymphocytes, Abs., Low - Last or Replicated | 0 | 0 | 0
  Ery. Mean Corpuscular Hemo., Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  Ery. Mean Corpuscular Hemo., Low - Any Abnormality | 0 | 0 | 1
  Ery. Mean Corpuscular Hemo., Low -Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  Ery. Mean Corpuscular Hemo., Low -Single, Not Last | 0 | 0 | 0
  Ery. Mean Corpuscular Hemo.,Low-Last or Replicated: number analyzed (Participants) | 80 | 53 | 72
  Ery. Mean Corpuscular Hemo.,Low-Last or Replicated | 0 | 0 | 1
  Neutrophils, Total, Abs., Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  Neutrophils, Total, Abs., Low - Any Abnormality | 1 | 1 | 0
  Neutrophils, Total, Abs., Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  Neutrophils, Total, Abs., Low - Single, Not Last | 1 | 0 | 0
  Neutrophils, Total, Abs., Low -Last or Replicated: number analyzed (Participants) | 80 | 53 | 72
  Neutrophils, Total, Abs., Low -Last or Replicated | 0 | 1 | 0
  Neutrophils, Total, Abs., High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  Neutrophils, Total, Abs., High - Any Abnormality | 2 | 0 | 2
  Neutrophils, Total, Abs., High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  Neutrophils, Total, Abs., High - Single, Not Last | 1 | 0 | 0
  Neutrophils, Total, Abs., High -Last or Replicated: number analyzed (Participants) | 80 | 53 | 72
  Neutrophils, Total, Abs., High -Last or Replicated | 1 | 0 | 2
  Platelets, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  Platelets, Low - Any Abnormality | 1 | 1 | 0
  Platelets, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  Platelets, Low - Single, Not Last | 0 | 0 | 0
  Platelets, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 72
  Platelets, Low - Last or Replicated | 1 | 1 | 0
  Platelets, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  Platelets, High - Any Abnormality | 1 | 0 | 0
  Platelets, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  Platelets, High - Single, Not Last | 0 | 0 | 0
  Platelets, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 72
  Platelets, High - Last or Replicated | 1 | 0 | 0
  Red Blood Cell Count, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  Red Blood Cell Count, Low - Any Abnormality | 3 | 1 | 1
  Red Blood Cell Count, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  Red Blood Cell Count, Low - Single, Not Last | 2 | 0 | 1
  Red Blood Cell Count, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 72
  Red Blood Cell Count, Low - Last or Replicated | 1 | 1 | 0
  White Blood Cell Count, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 72
  White Blood Cell Count, Low - Any Abnormality | 1 | 2 | 1
  White Blood Cell Count, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 72
  White Blood Cell Count, Low - Single, Not Last | 1 | 1 | 1
  White Blood Cell Count, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 72
  White Blood Cell Count, Low - Last or Replicated | 0 | 1 | 0

44. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Blood Chemistry Tests, in All Participants
Description: Clinical laboratory tests for blood chemistry parameters were performed and any marked abnormal values (High or Low) were based on Roche's predefined standard reference ranges. Marked laboratory abnormalities are presented according to COG3007 abnormality criteria: Single, Not Last = abnormality detected at a single assessment, but not at the last assessment; Last or Replicated = abnormality detected at the last assessment or replicated at one or more assessments. Not every laboratory abnormality qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy. SGOT/AST = serum glutamic oxaloacetic transaminase / aspartate aminotransferase
Time Frame: Predose at Baseline, Weeks 12 and 24, and at Early Termination and Unscheduled Visits (up to 36 weeks)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  Alkaline Phosphatase, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Alkaline Phosphatase, High - Any Abnormality | 0 | 0 | 1
  Alkaline Phosphatase, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Alkaline Phosphatase, High - Single, Not Last | 0 | 0 | 0
  Alkaline Phosphatase, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Alkaline Phosphatase, High - Last or Replicated | 0 | 0 | 1
  SGOT/AST, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  SGOT/AST, High - Any Abnormality | 0 | 1 | 0
  SGOT/AST, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  SGOT/AST, High - Single, Not Last | 0 | 0 | 0
  SGOT/AST, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  SGOT/AST, High - Last or Replicated | 0 | 1 | 0
  Bicarbonate, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Bicarbonate, Low - Any Abnormality | 4 | 1 | 2
  Bicarbonate, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Bicarbonate, Low - Single, Not Last | 0 | 0 | 1
  Bicarbonate, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Bicarbonate, Low - Last or Replicated | 4 | 1 | 1
  Bicarbonate, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Bicarbonate, High - Any Abnormality | 1 | 0 | 1
  Bicarbonate, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Bicarbonate, High - Single, Not Last | 0 | 0 | 0
  Bicarbonate, High - Last or Replicated: number analyzed (Participants) | 80 | 52 | 73
  Bicarbonate, High - Last or Replicated | 1 | 0 | 1
  Blood Urea Nitrogen, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Blood Urea Nitrogen, High - Any Abnormality | 2 | 3 | 3
  Blood Urea Nitrogen, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Blood Urea Nitrogen, High - Single, Not Last | 0 | 0 | 0
  Blood Urea Nitrogen, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Blood Urea Nitrogen, High - Last or Replicated | 2 | 3 | 3
  Calcium, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Calcium, Low - Any Abnormality | 2 | 0 | 2
  Calcium, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Calcium, Low - Single, Not Last | 1 | 0 | 1
  Calcium, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Calcium, Low - Last or Replicated | 1 | 0 | 1
  Chloride, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Chloride, Low - Any Abnormality | 3 | 1 | 0
  Chloride, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Chloride, Low - Single, Not Last | 2 | 1 | 0
  Chloride, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Chloride, Low - Last or Replicated | 1 | 0 | 0
  Cholesterol, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Cholesterol, High - Any Abnormality | 0 | 1 | 0
  Cholesterol, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Cholesterol, High - Single, Not Last | 0 | 0 | 0
  Cholesterol, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Cholesterol, High - Last or Replicated | 0 | 1 | 0
  Creatine Kinase, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Creatine Kinase, High - Any Abnormality | 3 | 0 | 1
  Creatine Kinase, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Creatine Kinase, High - Single, Not Last | 1 | 0 | 1
  Creatine Kinase, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Creatine Kinase, High - Last or Replicated | 2 | 0 | 0
  Creatinine, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Creatinine, High - Any Abnormality | 1 | 0 | 2
  Creatinine, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Creatinine, High - Single, Not Last | 0 | 0 | 0
  Creatinine, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Creatinine, High - Last or Replicated | 1 | 0 | 2
  Gamma Glutamyl Transferase, High-Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Gamma Glutamyl Transferase, High-Any Abnormality | 3 | 0 | 2
  Gamma Glutamyl Transferase, High-Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Gamma Glutamyl Transferase, High-Single, Not Last | 1 | 0 | 0
  Gamma Glutamyl Transferase,High-Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Gamma Glutamyl Transferase,High-Last or Replicated | 2 | 0 | 2
  Phosphorus, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Phosphorus, Low - Any Abnormality | 0 | 1 | 1
  Phosphorus, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Phosphorus, Low - Single, Not Last | 0 | 1 | 0
  Phosphorus, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Phosphorus, Low - Last or Replicated | 0 | 0 | 1
  Phosphorus, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Phosphorus, High - Any Abnormality | 3 | 0 | 1
  Phosphorus, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Phosphorus, High - Single, Not Last | 2 | 0 | 0
  Phosphorus, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Phosphorus, High - Last or Replicated | 1 | 0 | 1
  Potassium, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Potassium, High - Any Abnormality | 1 | 0 | 1
  Potassium, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Potassium, High - Single, Not Last | 0 | 0 | 1
  Potassium, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Potassium, High - Last or Replicated | 1 | 0 | 0
  Sodium, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Sodium, Low - Any Abnormality | 1 | 0 | 0
  Sodium, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Sodium, Low - Single, Not Last | 0 | 0 | 0
  Sodium, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Sodium, Low - Last or Replicated | 1 | 0 | 0
  Bilirubin, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Bilirubin, High - Any Abnormality | 0 | 0 | 1
  Bilirubin, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Bilirubin, High - Single, Not Last | 0 | 0 | 0
  Bilirubin, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Bilirubin, High - Last or Replicated | 0 | 0 | 1
  Protein, Total, Low - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  Protein, Total, Low - Any Abnormality | 0 | 0 | 1
  Protein, Total, Low - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  Protein, Total, Low - Single, Not Last | 0 | 0 | 0
  Protein, Total, Low - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  Protein, Total, Low - Last or Replicated | 0 | 0 | 1

45. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Coagulation Tests, in All Participants
Description: Clinical laboratory tests for coagulation parameters were performed and any marked abnormal values (High or Low) were based on Roche's predefined standard reference ranges. Marked laboratory abnormalities are presented according to COG3007 abnormality criteria: Single, Not Last = abnormality detected at a single assessment, but not at the last assessment; Last or Replicated = abnormality detected at the last assessment or replicated at one or more assessments. Not every laboratory abnormality qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy. aPTT = activated partial thromboplastin time; INR = International Normalized Ratio (prothrombin time)
Time Frame: Predose at Baseline, Weeks 12 and 24, and at Early Termination and Unscheduled Visits (up to 36 weeks)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 89 | 55 | 80
Participants
  INR, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  INR, High - Any Abnormality | 1 | 0 | 0
  INR, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  INR, High - Single, Not Last | 0 | 0 | 0
  INR, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  INR, High - Last or Replicated | 1 | 0 | 0
  aPTT, High - Any Abnormality: number analyzed (Participants) | 80 | 53 | 73
  aPTT, High - Any Abnormality | 5 | 1 | 1
  aPTT, High - Single, Not Last: number analyzed (Participants) | 80 | 53 | 73
  aPTT, High - Single, Not Last | 2 | 0 | 0
  aPTT, High - Last or Replicated: number analyzed (Participants) | 80 | 53 | 73
  aPTT, High - Last or Replicated | 3 | 1 | 1

46. Secondary Outcome: Number of Participants Who Tested Negative or Positive for Anti-Drug Antibodies Against Faricimab Over Time
Description: The number and percentage of participants who tested negative or positive for plasma anti-drug antibodies (ADA) to faricimab at baseline and at the study visits was tabulated, except for those who were randomized to treatment with ranibizumab in Arm A.
Time Frame: Baseline and Weeks 1, 4, 12, 16, 20, 24, 26, 28, 32, and 36
Population: Safety Population: all participants who had received at least one dose of the study drug, whether prematurely withdrawn from the study or not, grouped according to the actual treatment received. Analysis only included participants who were randomized to treatment with faricimab in Arms B and C.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
Number analyzed (Participants) | 0 | 55 | 80
Participants
  Baseline - ADA Negative: number analyzed (Participants) | 0 | 54 | 77
  Baseline - ADA Negative |  | 53 | 75
  Baseline - ADA Positive: number analyzed (Participants) | 0 | 54 | 77
  Baseline - ADA Positive |  | 1 | 2
  Week 1 - ADA Negative: number analyzed (Participants) | 0 | 52 | 68
  Week 1 - ADA Negative |  | 50 | 67
  Week 1 - ADA Positive: number analyzed (Participants) | 0 | 52 | 68
  Week 1 - ADA Positive |  | 2 | 1
  Week 4 - ADA Negative: number analyzed (Participants) | 0 | 53 | 76
  Week 4 - ADA Negative |  | 52 | 74
  Week 4 - ADA Positive: number analyzed (Participants) | 0 | 53 | 76
  Week 4 - ADA Positive |  | 1 | 2
  Week 12 - ADA Negative: number analyzed (Participants) | 0 | 51 | 71
  Week 12 - ADA Negative |  | 49 | 68
  Week 12 - ADA Positive: number analyzed (Participants) | 0 | 51 | 71
  Week 12 - ADA Positive |  | 2 | 3
  Week 16 - ADA Negative: number analyzed (Participants) | 0 | 1 | 1
  Week 16 - ADA Negative |  | 1 | 1
  Week 16 - ADA Positive: number analyzed (Participants) | 0 | 1 | 1
  Week 16 - ADA Positive |  | 0 | 0
  Week 20 - ADA Negative: number analyzed (Participants) | 0 | 52 | 70
  Week 20 - ADA Negative |  | 50 | 65
  Week 20 - ADA Positive: number analyzed (Participants) | 0 | 52 | 70
  Week 20 - ADA Positive |  | 2 | 5
  Week 24 - ADA Negative: number analyzed (Participants) | 0 | 49 | 64
  Week 24 - ADA Negative |  | 46 | 58
  Week 24 - ADA Positive: number analyzed (Participants) | 0 | 49 | 64
  Week 24 - ADA Positive |  | 3 | 6
  Week 26 - ADA Negative: number analyzed (Participants) | 0 | 2 | 5
  Week 26 - ADA Negative |  | 2 | 5
  Week 26 - ADA Positive: number analyzed (Participants) | 0 | 2 | 5
  Week 26 - ADA Positive |  | 0 | 0
  Week 28 - ADA Negative: number analyzed (Participants) | 0 | 6 | 7
  Week 28 - ADA Negative |  | 6 | 7
  Week 28 - ADA Positive: number analyzed (Participants) | 0 | 6 | 7
  Week 28 - ADA Positive |  | 0 | 0
  Week 32 - ADA Negative: number analyzed (Participants) | 0 | 5 | 5
  Week 32 - ADA Negative |  | 5 | 5
  Week 32 - ADA Positive: number analyzed (Participants) | 0 | 5 | 5
  Week 32 - ADA Positive |  | 0 | 0
  Week 36 - ADA Negative: number analyzed (Participants) | 0 | 36 | 53
  Week 36 - ADA Negative |  | 32 | 47
  Week 36 - ADA Positive: number analyzed (Participants) | 0 | 36 | 53
  Week 36 - ADA Positive |  | 4 | 6

ADVERSE EVENTS:
Time Frame: From Baseline until the final study visit (up to 36 weeks)
Arm/Group | Arm A: 0.3 mg Ranibizumab | Arm B: 1.5 mg Faricimab | Arm C: 6 mg Faricimab
All-Cause Mortality (participants affected / at risk) | 2/89 | 1/55 | 2/80
Serious Adverse Events (participants affected / at risk) | 9/89 | 7/55 | 8/80
Other Adverse Events (participants affected / at risk) | 48/89 | 31/55 | 45/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: 0.3 mg Ranibizumab (N=89) | Arm B: 1.5 mg Faricimab (N=55) | Arm C: 6 mg Faricimab (N=80)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Gangrene (Infections and infestations) | 1 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0
Hemiplegic migraine (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: 0.3 mg Ranibizumab (N=89) | Arm B: 1.5 mg Faricimab (N=55) | Arm C: 6 mg Faricimab (N=80)
Anaemia (Blood and lymphatic system disorders) | 9 | 1 | 5
Conjunctival haemorrhage (Eye disorders) | 7 | 2 | 8
Diabetic retinal oedema (Eye disorders) | 4 | 4 | 5
Dry eye (Eye disorders) | 2 | 0 | 4
Eye pain (Eye disorders) | 3 | 3 | 2
Retinal exudates (Eye disorders) | 1 | 4 | 3
Vision blurred (Eye disorders) | 2 | 3 | 2
Vitreous detachment (Eye disorders) | 3 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 4
Oedema peripheral (General disorders) | 3 | 2 | 4
Bronchitis (Infections and infestations) | 3 | 3 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 3 | 2
Nasopharyngitis (Infections and infestations) | 3 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 6
Urinary tract infection (Infections and infestations) | 6 | 4 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2
Hypertension (Vascular disorders) | 7 | 5 | 6
Cataract (Eye disorders) | 2 | 0 | 3
Eye pruritus (Eye disorders) | 3 | 1 | 1
Eyelid oedema (Eye disorders) | 0 | 2 | 0
Lacrimation increased (Eye disorders) | 3 | 0 | 1
Cataract subcapsular (Eye disorders) | 0 | 2 | 0
Vitreous haemorrhage (Eye disorders) | 3 | 0 | 0
Vitreous floaters (Eye disorders) | 2 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 3 | 0 | 0
Blood pressure increased (Investigations) | 3 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 3
Red blood cell sedimentation rate increased (Investigations) | 2 | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Headache (Nervous system disorders) | 2 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT02699450/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT02699450/SAP_001.pdf